CLINICAL TRIAL: NCT05587946
Title: The Effect of Virtual Reality Application Used During Endoscopy on Pain, Anxiety and Vital Signs: A Mixed Methods Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: İBRAHİM NAS (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, İBRAHİM NAS, Lecturer, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D. Tez
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Patient Relations, Nurse; Nurse's Role; Supportive Care
Keywords: Endoscopy; virtual reality; pain; anxiety; vital signs
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The Effect of Virtual Reality Application Used During Endoscopy on Pain, Anxiety and Vital Signs: A Mixed Methods Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/treatment (Experimental): 1. Implementation steps 1-4 of the Control Group will be done.
  2. The patient will be informed about the virtual reality application.
  3. The patient will be told that they can remove their glasses at any time and stop participating in the study.
  4. 2 minutes before the endoscopy process starts, the previously determined video will be started by putting on the Virtual Reality Glasses.
  5. Glasses will be worn from the beginning to the end of the procedure.
  6. The patient will be observed during the procedure. The data obtained during the observation will be noted.
  7. After the endoscopy procedure; "State Anxiety Scale", "Visual Comparison Scale" will be re-applied and vital signs will be measured and recorded in the Patient Follow-up Form.
  8. After the endoscopy procedure, patients will be given an interview appointment on the same day to collect the data of the qualitative part of the study.
  9. "Semi-Structured Interview Form" will be applied in the interview.
  Interventions: Other: Experimental group
- Control group (No Intervention): 1. Hands will be washed.
  2. The right patient will be determined, the procedure will be explained to the patient and permission will be obtained.
  3. A "Patient Identification Form" will be applied to the individual before the endoscopy procedure.
  4. Before the endoscopy procedure; "State Anxiety Scale" will be applied in the first 10 minutes, and "Visual Comparison Scale" will be applied in the first 5 minutes. Vital signs will be measured within the first 5 minutes and recorded on the Patient Follow-up Form. Then the individual will be taken to the endoscopy procedure.
  5. The patient will be observed during the procedure. The data obtained during the observation will be noted.
  6. After the endoscopy procedure; "State Anxiety Scale", "Visual Comparison Scale" will be applied again and vital signs will be measured and recorded in the Patient Follow-up Form.

INTERVENTIONS:
Other: Experimental group — In recent years, virtual reality has been widely used as a distraction practice in clinical medical care to relieve pain. Virtual reality is a method of viewing computer images to isolate the individual from real life for a while. Virtual reality glasses, consisting of a head-mounted display and glasses connected to a mobile phone, is a computer technology that creates a 3D environment. The virtual reality application, which was originally designed for entertainment purposes, started to be used in the medical field to reduce pain during invasive procedures in parallel with the developments in computer technologies. It is preferred in clinical practice as an easily accessible, non-invasive and inexpensive method.
  Other Names: Girişim grubu
  Arms: Intervention/treatment

SUMMARY:
In this study, the effect of virtual reality application used during upper gastrointestinal endoscopy on pain, anxiety and vital signs will be investigated. The research will be conducted as a mixed methods research including quantitative and qualitative methods. The exploratory sequence mixed design model, one of the mixed method designs, will be used in the research.

DETAILED DESCRIPTION:
Objective: In this study, the effect of virtual reality application used during upper gastrointestinal endoscopy on pain, anxiety and vital signs will be investigated. The research will be conducted as a mixed methods research including quantitative and qualitative methods. The exploratory sequence mixed design model, one of the mixed method designs, will be used in the research.

The research was carried out in the endoscopy unit of a university hospital in Van between November 2022 and March 2023. This research, in which an exploratory sequential mixed design was used, consists of two stages. In the research, the quantitative phase, in which a pretest-posttest design, randomized controlled, experimental method was used, was completed with 75 patients, and the qualitative phase, in which the phenomenological/phenomenological design was used, was completed with 19 patients. Patient introduction form, state anxiety scale, pain visual comparison scale, patient follow-up form and semi-structured interview form were used to collect data. IBM SPSS V23 program (quantitative) and inductive qualitative content analysis (qualitative) were used to analyze the data.

ELIGIBILITY:
Criteria:

Inclusion criteria:

Inclusion criteria for the quantitative study;

* 18 years and older,
* who can read and write Turkish,
* without mental problems,
* Having no vision, hearing or perception problems,
* Diagnostic endoscopy was performed,
* No sedation before and during the procedure
* who volunteered to participate in the study,
* Those who have not taken analgesics in the last 8 hours

Qualitative research inclusion criteria;

* in the experimental group,
* who volunteered to participate in the research

Exclusion Criteria:

Exclusion criteria from quantitative section research;

* sedation applied,
* who want to withdraw from the study,
* Patients using analgesics or anti-anxiety medications before and during the procedure

Exclusion criteria from qualitative departmental research;

• Those in the control group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety state before endoscopy | Anxiety state reported within the first 10 minutes before the endoscopy procedure
  The statements in the state anxiety scale were answered as "not at all", "a little", "a lot" and "totally" according to the feelings of the person. A total score of 20-80 is obtained from the scale. A low score indicates a low level of anxiety, and a high one indicates a high level of anxiety. The score obtained from the scale, on the other hand, indicates mild anxiety between 20-39, moderate anxiety between 40-59 and severe anxiety between 60-80.
Pain intensity before endoscopy | Pain intensity reported within the first 5 minutes prior to the endoscopy procedure
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst Pain
Heart rate before the endoscopy procedure | Just before the endoscopy procedure
  60 to 100 beats per minute is normal.
Blood pressure before the endoscopy procedure | Just before the endoscopy procedure
  90/60 mm Hg to 120/80 mm/Hg is normal.
Respiration rate before the endoscopy procedure | Just before the endoscopy procedure
  12 to 20 breaths per minute is normal.
Body temperature before the endoscopy procedure | Just before the endoscopy procedure
  Normal Body temperature; 36 to 37-5 degrees is normal.
Oxygen saturation (SpO2) before the endoscopy procedure | Just before the endoscopy procedure
  Normal oxygen saturation usually ranges from 95% to 100%.
Oxygen saturation (SpO2) after endoscopy procedure | within first 5 minutes after endoscopy procedure
  Normal oxygen saturation usually ranges from 95% to 100%.
Body temperature after endoscopy procedure | within first 5 minutes after endoscopy procedure
  Normal Body temperature; 36 to 37-5 degrees is normal.
Respiration rate after endoscopy procedure | Respiratory rate/minute reported in the first 5 minutes after the endoscopy procedure
  12 to 20 breaths per minute is normal.
Blood pressure after the endoscopy procedure | within first 5 minutes after the endoscopy procedure
  90/60 mm Hg to 120/80 mm/Hg is normal.
Heart rate after the endoscopy procedure | Heart rate per minute reported in the first 5 minutes after the endoscopy procedure
  60 to 100 beats per minute is normal.
Post-endoscopy pain | Pain severity reported in the first 5 minutes after the endoscopy procedure
  Pain severity assessment with Visual Assessment Scale (VAS) Score: 0-10; 0- No Pain, 10- Worst Pain
Post-endoscopy anxiety state | Anxiety state reported within the first 10 minutes after the endoscopy procedure
  The statements in the state anxiety scale were answered as "not at all", "a little", "a lot" and "totally" according to the feelings of the person. A total score of 20-80 is obtained from the scale. A low score indicates a low level of anxiety, and a high one indicates a high level of anxiety. The score obtained from the scale, on the other hand, indicates mild anxiety between 20-39, moderate anxiety between 40-59 and severe anxiety between 60-80.

SECONDARY OUTCOMES:
Patient opinions on endoscopy | Two hours after endoscopy
  General thoughts of the patient about endoscopy
Patient opinions on virtual reality glasses and its application | Two hours after endoscopy
  General thoughts of the patient about the use of virtual reality glasses during endoscopy
Patient opinions on the effect of virtual reality application on pain | Two hours after endoscopy
  Patient opinions on the effect of virtual reality application on pain
Patient opinions on the effect of virtual reality application on anxiety | Two hours after endoscopy
  Patient opinions on the effect of virtual reality application on anxiety

CONTACTS AND LOCATIONS:
Overall Officials: GÜLAY İPEK ÇOBAN, Prof.Dr., Principal Investigator — Ataturk University
Locations (1):
- Van Yüzüncü Yıl University, Faculty of Health Sciences, Department of Nursing, Van, Turkey, Van, Turkey (Türkiye)